CLINICAL TRIAL: NCT00628225
Title: Smoking Cessation in Patients With COPD (SMOCC) in General Practice
Acronym: SMOCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Collaborators: The Netherlands Asthma Foundation (Other); Pharmacia (Industry); GlaxoSmithKline (Industry)
Responsible Party: Dr. A. Jacobs, Radboud University Nijmegen Medical Centre
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zonmw22000039; GlaxoSmithKline ZYB40023; Pharmacia HK/jh/00013; Dutch Asthma Found. 3.4.98.47
Record Dates: First submitted 2008-02-25; First posted 2008-03-04 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Smoking cessation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation | interventions — Counseling; Nicotine Replacement Therapy; Bupropion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Usual Care
- 2 (Experimental): Multifacetted smoking cessation intervention (aimed at professional (training and education) and at patients (counseling + nicotine replacement)
  Interventions: Behavioral: Counseling and Nicotine replacement (CN)
- 3 (Experimental): Multifacetted smoking cessation intervention (aimed at professional (training and education) and at patients (counseling + nicotine replacement + bupropion-SR)
  Interventions: Behavioral: Counseling, Nicotine replacement and Bupropion (CNB)

INTERVENTIONS:
Behavioral: Counseling and Nicotine replacement (CN) — Professionals in general practice received a central training (4 hours) about smoking, smoking cessation and COPD. They received materials (leaflet, video, smoking cessation protocol and informationfolder). Moreover, professionals received a maximum of 4 practice visits from an outreach visitor. General practitioners were encouraged to advise nicotine replacement.
  Smoking COPD patients received smoking cessation counseling and were advised to use nicotine replacement.
  Arms: 2
Behavioral: Counseling, Nicotine replacement and Bupropion (CNB) — Professionals in general practice received a central training (4 hours) about smoking, smoking cessation and COPD. They received materials (leaflet, video, smoking cessation protocol and informationfolder). Moreover, professionals received a maximum of 4 practice visits from an outreach visitor. The general practitioner was encouraged to advice the patients to use both nicotine replacements and Bupropion-SR.
  Smoking COPD patients received smoking cessation counseling and were advised to use nicotine replacement and Bupropion-SR.
  Other Names: Bupropion-SR (Zyban)
  Arms: 3

SUMMARY:
Background: Smoking cessation is the key element in the treatment of patients with Chronic Obstructive Pulmonary Disease (COPD). The role of the general practice in assisting these patients with successful quitting smoking was suboptimal. Therefore we evaluated the effectiveness of two smoking cessation programs (counseling and nicotine replacement) for smokers with COPD in routine general practice, one with (CNB) and one without (CN) the combination with bupropion-SR, compared to usual care (UC) and explored the role of COPD symptoms in successful smoking cessation.

Method: RCT with 667 patients with COPD, 68 general practices were randomly allocated. The usual care group (UC) consisted of 148 patients (22 practices), the first intervention group (counseling plus nicotine replacement (CN) of 243 patients (21 practices) and the second intervention group of 276 patients (25 practices. Main outcome measure was (biochemically verified) point prevalence.

ELIGIBILITY:
Inclusion Criteria:

A software program using Anatomical Therapeutical Chemical (ATC) prescription codes and International Classification of Primary Care (ICPC) diagnosis codes selected potential patients with COPD. Criteria: age >35 years and a diagnosis recorded as COPD or as ICPC code R95/96, or a prescription of at least three times of bronchodilators (ATC code R03a/bc) and/or prescription of at least two times of inhaled anti-inflammatory medication in the past year (ATC code R03). General practitioners (GPs) had to confirm the diagnosis of the selection. Patients were eligible to participate if they met the following criteria:

* Current smoking
* Suffering from COPD according to the GP's diagnosis
* In command of the Dutch language.

Exclusion Criteria:

* Too ill
* Under control of a chest physician
* Serious physical or psychological comorbidity

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2000-03; Primary Completion 2002-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Smoking cessation (point prevalence, both self reported as biochemical verified) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Annelies E Jacobs, PHD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Result] Hilberink SR, Jacobs JE, Schlosser M, Grol RP, de Vries H. Characteristics of patients with COPD in three motivational stages related to smoking cessation. Patient Educ Couns. 2006 Jun;61(3):449-57. doi: 10.1016/j.pec.2005.05.012. Epub 2005 Sep 12. PMID 16157462
- [Result] Hilberink SR, Jacobs JE, Bottema BJ, de Vries H, Grol RP. Smoking cessation in patients with COPD in daily general practice (SMOCC): six months' results. Prev Med. 2005 Nov-Dec;41(5-6):822-7. doi: 10.1016/j.ypmed.2005.08.003. Epub 2005 Oct 3. PMID 16203030
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Hilberink SR, Jacobs JE, Breteler MH, de Vries H, Grol RP. General practice counseling for patients with chronic obstructive pulmonary disease to quit smoking: impact after 1 year of two complex interventions. Patient Educ Couns. 2011 Apr;83(1):120-4. doi: 10.1016/j.pec.2010.04.009. Epub 2010 Apr 28. PMID 20430565